CLINICAL TRIAL: NCT04091763
Title: Sclerotherapy With Polidocanol Foam Versus Rubber Band Ligation in the Treatment of First, Second and Third-Grade Hemorrhoidal Disease: a Randomized, Controlled Trial
Brief Title: Polidocanol Foam Versus Rubber Band Ligation in the Treatment of Hemorrhoidal Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Paulo Sérgio Durão Salgueiro, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209117311
Record Dates: First submitted 2019-09-04; First posted 2019-09-17 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Hemorrhoids, Internal
Keywords: Sclerotherapy; Rubber band ligation; Polidocanol foam; Hemorrhoidal disease
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either rubber band ligation or sclerotherapy with polidocanol foam, stratified by grade of hemorrhoidal disease
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polidocanol foam sclerotherapy (Experimental): 1. Preparation of the polidocanol foam according to Tessari technique immediately before application (so that the "microbubbles" of the foam did not disintegrate);
  2. Application according to the Blanchard technique (Fig. 2) through a disposable transparent anoscope, with the patient in jackknife position, using a 20mL disposable syringe of the mixture (polidocanol + air) and a reusable 10 cm syringe extender adapted to an intravenous needle;
  3. Patients treated in a maximum of 3 sessions at 3 weeks intervals;
  4. Maximum dose per treatment session of 20mL of mixture of 4mL of polidocanol 3% with 16mL of air;
  5. In each session more than one hemorrhoid cushion could be treated.
  Interventions: Drug: Polidocanol Injectable Foam
- Rubber band ligation (Experimental): 1. Use of reusable metal ligation device connected to a vacuum system (McGown suction method) to apply the rubber bands above the dentated line through a disposable transparent anoscope with the patient in jackknife position;
  2. A maximum of 3 sessions of ligation at 3-week intervals were performed;
  3. More than 1 band per session could be applied.
  Interventions: Device: Rubber band ligation

INTERVENTIONS:
Drug: Polidocanol Injectable Foam — Two distinct periods were considered: intervention and follow-up. During the intervention period patients were observed at 3-week intervals (minimum of 3 weeks and maximum of 9 weeks depending on the number of instrumental treatments performed). The required number of sessions of any of the office-based treatments (maximum of 3 sessions) was determined by clinical and anoscopy response (if after the treatment the participant scored zero points in the Sodergren scale or the anoscopy did not reveal significant hemorrhoidal disease, there was no place for additional instrumental therapy and the patient started the follow-up period.
  If there was therapeutic failure at the end of the third session or if there was a significant complication (moderate or severe) the patient's participation in the study ended and he was referred for treatment with other type of office-based procedure or surgery.
  Arms: Polidocanol foam sclerotherapy
Device: Rubber band ligation — Two distinct periods were considered: intervention and follow-up. During the intervention period patients were observed at 3-week intervals (minimum of 3 weeks and maximum of 9 weeks depending on the number of instrumental treatments performed). The required number of sessions of any of the office-based treatments (maximum of 3 sessions) was determined by clinical and anoscopy response (if after the treatment the participant scored zero points in the Sodergren scale or the anoscopy did not reveal significant hemorrhoidal disease, there was no place for additional instrumental therapy and the patient started the follow-up period.
  If there was therapeutic failure at the end of the third session or if there was a significant complication (moderate or severe) the patient's participation in the study ended and he was referred for treatment with other type of office-based procedure or surgery.
  Arms: Rubber band ligation

SUMMARY:
Background: Hemorrhoidal disease is a common benign condition seen frequently in clinical settings. Rubber band ligation and sclerotherapy have proven to be the office-based procedures of choice in hemorrhoidal disease, with various studies reporting rubber band ligation as being more effective but also more painful and bleeding prone than sclerotherapy with liquid polidocanol. However, there are no studies comparing rubber band ligation and sclerotherapy with polidocanol foam, a new type of sclerosant agent that has already proved to be more effective and safer than liquid polidocanol in grade I hemorrhoidal disease.

The present study was designed to establish the clinical effectiveness and safety of sclerotherapy with polidocanol foam compared with rubber band ligation.

Methods: This randomized controlled trial includes patients with symptomatic hemorrhoidal disease grades I to III. The participants were randomly assigned (in a 1:1 ratio) to either rubber band ligation or sclerotherapy with polidocanol foam, stratified by grade of hemorrhoidal disease. During the intervention period the patients are submitted to one of the office-based procedures and, afterwards, in the follow-up period, evaluated every three months for a total period of one year.

The efficacy outcomes include symptom resolution, number of treatment sessions needed to achieve therapeutic success and evolution of hemorrhoidal disease grade in the intervention period and, during follow-up, recurrence incidence. Primary safety outcomes include the occurrence of any complication related to the office-based procedures.

DETAILED DESCRIPTION:
INTRODUCTION Hemorrhoids are normal vascular structures in the anal canal, arising from a cushion of dilated arteriovenous channels and connective tissues, that drains into the superior and inferior hemorrhoidal veins. Their main function is to maintain anal continence, serve as a protection for the anal sphincters during the act of defecation and have a sensory function, allowing to differentiate liquids, solids or gases and to signal defecation.

The hemorrhoidal disease develops when the supporting tissues of hemorrhoidal cushions deteriorate due to various processes: abnormal venous dilation, vascular thrombosis, degenerative processes of collagen and fibroelastic tissue, distortion and rupture of anal subepithelial muscle, hyperperfusion of the hemorrhoidal plexus, inflammatory phenomena and hormonal changes (typical of pregnancy).

Hemorrhoidal disease occurs frequently in the adult population and a considerable number of patients are asymptomatic. Both sexes are similarly affected. The peak incidence occurs between 45-65 years, being rare before the age of 20.

Classification of hemorrhoidal disease corresponds to its position relative to the dentate line. External hemorrhoids are located below the dentate line and are covered by modified squamous epithelium, being richly innervated and therefore painful when there is associated thrombosis. On the contrary, internal hemorrhoids lie above the dentate line. Internal hemorrhoids are further classified based on their appearance and degree of prolapse according to the Goligher classification: grade I, without prolapse (they have the potential to bleed but are not visualized without the aid of an anoscope); grade II, prolapsed with defecation, but reduced spontaneously; grade III, prolapse with defecation requiring manual reduction and grade IV, prolapsed and non-reducible.

Since hemorrhoidal disease is a benign pathology, its treatment should be guided by the symptoms and the impact of the disease on quality of life. A prospective study by Pucher et al. developed and validated the Sodergren scale, which is based on a set of symptoms to assess the severity of hemorrhoidal disease. This scale can be used to assess the efficacy of treatment of haemorrhoids and the comparison of trials, consequently it is helpful in the choice of the best therapeutic option.

Treatment of hemorrhoidal disease can be divided into conservative measures, office-based procedures and surgical treatments.

First line therapy should be conservative and includes a set of lifestyle changes, dietary changes, laxative medication and phlebotonic and/or topical anti-inflammatory drugs. These measures produce beneficial effects and should be implemented in every grades of hemorrhoidal disease or in patients undergoing instrumental or surgical treatment.

The instrumental office-based treatment is usually indicated for hemorrhoidal disease grade I and II, thought it can also be used in grade III hemorrhoidal disease. It is aimed at decreasing hemorrhoidal vascularization, reducing redundant tissue and increasing hemorrhoidal rectal wall fixation to minimize prolapse. It includes rubber band ligation, sclerotherapy (liquid and foam agents), infrared photocoagulation, cryotherapy and radiofrequency ablation.

Rubber band ligation is the most commonly performed procedure in the office and is indicated for grade II and III internal hemorrhoids and works by causing hemorrhoid tissue necrosis and its fixation to the rectal mucosa. Complications associated with rubber band ligation include bleeding (ranging from mild to severe), pain, urinary symptoms, priapism, vagal symptoms, hemorrhoidal thrombosis, sepsis, fistulation or even death. Hemorrhage and pain are among the most frequent. Cumulatively, a success rate of 80% is observed with rubber band ligation.

Hemorrhoidal sclerosis is a procedure commonly used to treat grade I and II hemorrhoidal disease. It has also been used in internal grade III hemorrhoids, although in these cases there is little scientific evidence supporting its efficacy. In this technique a needle is introduced through an endoscope or anoscope and the sclerosing agent is injected into the hemorrhoid above the dentated line - Blanchard technique.

There are a variety of sclerosing agents such as 5% phenol in vegetable oil, quinine, tetradecyl sodium sulfate, sodium morphate or potassium aluminum sulfate and tannic acid (ALTA). More recently, a new sclerosing substance, polidocanol, a non-ionic detergent consisting of two components, a polar hydrophilic chain and a non-polar hydrophobic, started to be employed in the treatment of hemorrhoidal disease. The experience of its use in sclerotherapy comes mainly from the treatment of varicose veins and it can be used in its liquid or foam form. Several studies reported the efficacy of the use of sclerotherapy with liquid polidocanol in hemorrhoidal disease; it is considered a sclerosing agent with anesthetic properties, well tolerated, with low necrotic potential and a very promising agent for the treatment of grade I hemorrhoidal disease. The foam formation is based on the Tessari technique which uses a device that combines two syringes and a three-way tap in which the polidocanol is mixed with air under mechanical force ("Tourbillon technique"). This formulation allows for greater efficacy and use of lower doses of sclerosing agent since the volume will be greatly increased and hence also the area of contact with the vascular endothelium where the drug will exert its sclerosing action. The use of polidocanol foam in the treatment of varicose veins is safe and effective and has been shown to be superior to the use of liquid polidocanol. Its use is not indicated in cases of acute thromboembolism and allergy to polidocanol.

There is only one study showing the superiority of polidocanol foam compared to its liquid formulation in the treatment of grade I hemorrhoidal disease. In a recently published non-controlled study, 2000 patients with hemorrhoidal disease grades I to IV were treated with polidocanol foam and the authors concluded that this therapy was very successful, with 98% of the patients reporting satisfaction regarding bleeding control and prolapse reduction. Complications were rare and usually minor. There's a lack of studies comparing it with other ablative techniques.

The most common complications of sclerotherapy include mild anal discomfort and bleeding. However, the bleeding risk is lower compared to that observed with rubber band ligation. Rare complications include erectile dysfunction, mucosal ulceration, necrosis, prostatic abscess, retroperitoneal sepsis and transient bacteremia. Sclerotherapy is a valid alternative for the treatment of patients whose hemorrhage is the main symptom and where conservative therapy has not been effective, as well as for patients on anticoagulant medication, and for cirrhotic or immunocompromised patients.

There have been no comparative studies between polidocanol foam sclerotherapy and rubber band ligation.

With the present study, the investigators aim to fill a gap in the literature by evaluating the safety and efficacy in the treatment of hemorrhoidal disease with the seemingly most effective non-surgical office-based methods (rubber band ligation and sclerotherapy with polidocanol foam).

METHODS PARTICIPANTS AND ETHICAL ASPECTS Are included patients referred to proctologic consultation of Centro Hospitalar Universitário do Porto (CHUP) older than 18 years with symptomatic hemorrhoidal disease grade I, II and III (Goligher's classification) refractory to conservative management (dietary modification, intestinal transit modifiers, topical and phlebotonic medications) for a period of no less than 4 weeks. All participants must have prior endoscopic study, at least recto-sigmoidoscopy, or complete colonoscopy if they are older than 50 years or younger with family history of colorectal cancer, colon adenomas, or suspected inflammatory bowel disease.

The study was approved by the ethics committee of CHUP. All the participants enrolled sign an informed consent.

STATISTICAL ANALYSIS Sample size was determined considering a power of 80% (type II error ß of 20%) and significance level α of 5% (type I error). The required number in each treatment was 44 patients. In order to safeguard against potential drop-outs, a sample size of 120 (60+60) patients was considered.

It was generated a 1:1 randomization sequence, stratified by for the degree of hemorrhoidal disease (Goligher's classification), to assign participants to each one of the therapeutic arms either sclerotherapy with polidocanol foam or rubber band ligation.

Since the two office-based therapies under study have completely different techniques and procedures, it is not possible to blind either the patient or the clinician who apply the treatment. Therefore, an open label study is being conducted.

VISITS AND DATA COLLECTION Demographic data such as age, sex, body mass index (BMI) are collected. In the first visit informed consent and an information brochure explaining the study and adequate dietary and behavioral care is provided.

For purposes of evaluating efficacy and safety, two distinct periods were considered: intervention and follow-up.

During the intervention period, when office-based treatments are performed, patients are observed at 3-week intervals (minimum of 3 weeks and maximum of 9 weeks depending on the number of instrumental treatments performed) and, during follow-up period, every 3 months, 3 weeks after the last session of treatment to evaluate recurrence of hemorrhoidal disease (maximum 1 year; 4 visits).

At all visits, a proctologic examination with anoscopy is performed and clinical evaluation is carried out by filling the Sodergren's scale of symptoms. The severity of bleeding is also evaluated.

INTERVENTION PERIOD AND TECHNICAL ASPECTS The required number of sessions of any of the office-based treatments (maximum of 3 sessions) is determined by clinical and anoscopy response i.e., if 3 weeks after the previous treatment the participant scores zero points in the Sodergren scale and has bleeding grade ≤1 or the anoscopy doesn't reveal significant hemorrhoidal disease, there is no place for additional instrumental therapy and the patient starts the follow-up period.

If there is therapeutic failure (participants that, at the end of three sessions of instrumental treatment, aggravate or maintain the initial Sodergren score and bleeding grade) or if there is a significant complication (moderate or severe) the patient's participation in the study ends and he is referred for treatment with other type of office-based procedure or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to proctologic consultation of Centro Hospitalar Universitário do Porto (CHUP) older than 18 years;
* Clinical diagnosis of hemorrhoidal disease grade I, II and III (Goligher's classification);
* Refractory to conservative management (dietary modification, intestinal transit modifiers, topical and phlebotonic medications) for a period of no less than 4 weeks.

Exclusion Criteria:

* Hepatic cirrhosis;
* Pregnant or breast-feeding women;
* Known allergy to polidocanol
* Another perianal disease that can cause symptoms similar to hemorrhoidal disease;
* Concomitant presence of external hemorrhoidal disease and/or hemorrhoidal thrombosis;
* Office-based or surgical treatment for hemorrhoids within 6 months prior to inclusion;
* Antiplatelet or hypocoagulant medication;
* Inherited bleeding disorders;
* Immunosuppressive states ;
* Inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome (therapeutic success) | Three to nine weeks (depending on the number of instrumental treatments performed)
  Achievement of therapeutic success. Classified as:
  1. Complete (Sodergren score = 0 and bleeding grade ≤ 1);
  2. Partial (Sodergren score> 0 and bleeding grade > 1 but with improvement over initial score);
  3. Therapeutic failure (participants that, at the end of three sessions of instrumental treatment, aggravated or maintained the initial Sodergren score and bleeding grade).
Efficacy outcome (recurrence) | One year (after the last office-based procedure)
  Recurrence of hemorrhoidal disease during the follow-up period (only for patients who have had some degree of therapeutic success). Classified as:
  1. Mild (Sodergren score and bleeding grade higher than the evaluation at the beginning of the follow-up period but lower than the initial ones without the need for instrumental or surgical intervention);
  2. Severe (Sodergren score and degree of hemorrhage ≥ the initial one requiring instrumental or surgical intervention).
Safety outcome | Three to nine weeks (depending on the number of instrumental treatments performed)
  Complications resulting from the office-based procedures are recorded and classified as:
  1. Mild (e.g. pain/discomfort; pruritus; bright red blood on toilet paper/cleaning pad, hemorrhoidal thrombosis requiring only medical treatment);
  2. Moderate (e.g. external hemorrhoidal thrombosis requiring surgical intervention; bright red blood that drips in the toilet or clot expulsion not requiring blood transfusion, urgent hemostasis or urgent surgery): obliges the participant to be withdrawn from the study but do not endanger the patient's life or leave long term sequelae;
  3. Severe (e.g. sepsis; Fournier's gangrene; perineal abscess; bleeding with hemodynamic instability, transfusional need or urgent surgery; sexual impotence in man): obliges the participant to be withdrawn from the study and put the patient's life at risk or implies long-term sequelae.

SECONDARY OUTCOMES:
Efficacy outcome (number of sessions) | Three to nine weeks (depending on the number of instrumental treatments performed)
  Number of instrumental treatment sessions required to achieve therapeutic success.
Efficacy outcome (Goligher grade) | Three to nine weeks (depending on the number of instrumental treatments performed)
  Evolution of the grade of hemorrhoidal disease (Goligher's classification).

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Salgueiro, MD, Principal Investigator — Gastrenterologist
Locations (1):
- Centro Hospitalar Universitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sneider EB, Maykel JA. Diagnosis and management of symptomatic hemorrhoids. Surg Clin North Am. 2010 Feb;90(1):17-32, Table of Contents. doi: 10.1016/j.suc.2009.10.005. PMID 20109630
- [Background] Lohsiriwat V. Hemorrhoids: from basic pathophysiology to clinical management. World J Gastroenterol. 2012 May 7;18(17):2009-17. doi: 10.3748/wjg.v18.i17.2009. PMID 22563187
- [Background] Lohsiriwat V. Approach to hemorrhoids. Curr Gastroenterol Rep. 2013 Jul;15(7):332. doi: 10.1007/s11894-013-0332-6. PMID 23715885
- [Background] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Background] Johanson JF, Sonnenberg A. The prevalence of hemorrhoids and chronic constipation. An epidemiologic study. Gastroenterology. 1990 Feb;98(2):380-6. doi: 10.1016/0016-5085(90)90828-o. PMID 2295392
- [Background] Qureshi WA. Office management of hemorrhoids. Am J Gastroenterol. 2018 Jun;113(6):795-798. doi: 10.1038/s41395-018-0020-0. No abstract available. PMID 29487411
- [Background] Pucher PH, Qurashi M, Howell AM, Faiz O, Ziprin P, Darzi A, Sodergren MH. Development and validation of a symptom-based severity score for haemorrhoidal disease: the Sodergren score. Colorectal Dis. 2015 Jul;17(7):612-8. doi: 10.1111/codi.12903. PMID 25603811
- [Background] Sun Z, Migaly J. Review of Hemorrhoid Disease: Presentation and Management. Clin Colon Rectal Surg. 2016 Mar;29(1):22-9. doi: 10.1055/s-0035-1568144. PMID 26929748
- [Background] Hollingshead JR, Phillips RK. Haemorrhoids: modern diagnosis and treatment. Postgrad Med J. 2016 Jan;92(1083):4-8. doi: 10.1136/postgradmedj-2015-133328. Epub 2015 Nov 11. PMID 26561592
- [Background] Sandler RS, Peery AF. Rethinking What We Know About Hemorrhoids. Clin Gastroenterol Hepatol. 2019 Jan;17(1):8-15. doi: 10.1016/j.cgh.2018.03.020. Epub 2018 Mar 27. PMID 29601902
- [Background] Ganz RA. The evaluation and treatment of hemorrhoids: a guide for the gastroenterologist. Clin Gastroenterol Hepatol. 2013 Jun;11(6):593-603. doi: 10.1016/j.cgh.2012.12.020. Epub 2013 Jan 16. No abstract available. PMID 23333220
- [Background] Albuquerque A. Rubber band ligation of hemorrhoids: A guide for complications. World J Gastrointest Surg. 2016 Sep 27;8(9):614-620. doi: 10.4240/wjgs.v8.i9.614. PMID 27721924
- [Background] Cocorullo G, Tutino R, Falco N, Licari L, Orlando G, Fontana T, Raspanti C, Salamone G, Scerrino G, Gallo G, Trompetto M, Gulotta G. The non-surgical management for hemorrhoidal disease. A systematic review. G Chir. 2017 Jan-Feb;38(1):5-14. doi: 10.11138/gchir/2017.38.1.005. PMID 28460197
- [Background] Iyer VS, Shrier I, Gordon PH. Long-term outcome of rubber band ligation for symptomatic primary and recurrent internal hemorrhoids. Dis Colon Rectum. 2004 Aug;47(8):1364-70. doi: 10.1007/s10350-004-0591-2. PMID 15484351
- [Background] Acheson AG, Scholefield JH. Management of haemorrhoids. BMJ. 2008 Feb 16;336(7640):380-3. doi: 10.1136/bmj.39465.674745.80. No abstract available. PMID 18276714
- [Background] Brown SR. Haemorrhoids: an update on management. Ther Adv Chronic Dis. 2017 Oct;8(10):141-147. doi: 10.1177/2040622317713957. Epub 2017 Jun 21. PMID 28989595
- [Background] Hachiro Y, Kunimoto M, Abe T, Kitada M, Ebisawa Y. Aluminum potassium sulfate and tannic acid (ALTA) injection as the mainstay of treatment for internal hemorrhoids. Surg Today. 2011 Jun;41(6):806-9. doi: 10.1007/s00595-010-4386-x. Epub 2011 May 28. PMID 21626327
- [Background] Herold A, Dietrich J, Aitchison R. Intra-anal Iferanserin 10 mg BID for hemorrhoid disease: a prospective, randomized, double-blind, placebo-controlled trial. Clin Ther. 2012 Feb;34(2):329-40. doi: 10.1016/j.clinthera.2011.12.012. Epub 2012 Jan 11. PMID 22244049
- [Background] Hussar DA, Stevenson T. New drugs: Denosumab, dienogest/estradiol valerate, and polidocanol. J Am Pharm Assoc (2003). 2010 Sep-Oct;50(5):658-62. doi: 10.1331/JAPhA.2010.10536. No abstract available. PMID 20833626
- [Background] Yuksel BC, Armagan H, Berkem H, Yildiz Y, Ozel H, Hengirmen S. Conservative management of hemorrhoids: a comparison of venotonic flavonoid micronized purified flavonoid fraction (MPFF) and sclerotherapy. Surg Today. 2008;38(2):123-9. doi: 10.1007/s00595-007-3582-9. Epub 2008 Feb 1. PMID 18239868
- [Background] Tessari L, Cavezzi A, Frullini A. Preliminary experience with a new sclerosing foam in the treatment of varicose veins. Dermatol Surg. 2001 Jan;27(1):58-60. PMID 11231246
- [Background] Cavezzi A, Tessari L. Foam sclerotherapy techniques: different gases and methods of preparation, catheter versus direct injection. Phlebology. 2009 Dec;24(6):247-51. doi: 10.1258/phleb.2009.009061. PMID 19952380
- [Background] Nastasa V, Samaras K, Ampatzidis Ch, Karapantsios TD, Trelles MA, Moreno-Moraga J, Smarandache A, Pascu ML. Properties of polidocanol foam in view of its use in sclerotherapy. Int J Pharm. 2015 Jan 30;478(2):588-96. doi: 10.1016/j.ijpharm.2014.11.056. Epub 2014 Nov 26. PMID 25433198
- [Background] Hamel-Desnos C, Desnos P, Wollmann JC, Ouvry P, Mako S, Allaert FA. Evaluation of the efficacy of polidocanol in the form of foam compared with liquid form in sclerotherapy of the greater saphenous vein: initial results. Dermatol Surg. 2003 Dec;29(12):1170-5; discussion 1175. doi: 10.1111/j.1524-4725.2003.29398.x. PMID 14725657
- [Background] Jia X, Mowatt G, Burr JM, Cassar K, Cook J, Fraser C. Systematic review of foam sclerotherapy for varicose veins. Br J Surg. 2007 Aug;94(8):925-36. doi: 10.1002/bjs.5891. PMID 17636511
- [Background] Moser KH, Mosch C, Walgenbach M, Bussen DG, Kirsch J, Joos AK, Gliem P, Sauerland S. Efficacy and safety of sclerotherapy with polidocanol foam in comparison with fluid sclerosant in the treatment of first-grade haemorrhoidal disease: a randomised, controlled, single-blind, multicentre trial. Int J Colorectal Dis. 2013 Oct;28(10):1439-47. doi: 10.1007/s00384-013-1729-2. Epub 2013 Jun 18. PMID 23775099
- [Background] Fernandes V, Fonseca J. Polidocanol Foam Injected at High Doses with Intravenous Needle: The (Almost) Perfect Treatment of Symptomatic Internal Hemorrhoids. GE Port J Gastroenterol. 2019 May;26(3):169-175. doi: 10.1159/000492202. Epub 2018 Aug 31. PMID 31192285
- [Background] Scaglia M, Delaini GG, Destefano I, Hulten L. Injection treatment of hemorrhoids in patients with acquired immunodeficiency syndrome. Dis Colon Rectum. 2001 Mar;44(3):401-4. doi: 10.1007/BF02234740. PMID 11289287
- [Background] MacRae HM, McLeod RS. Comparison of hemorrhoidal treatment modalities. A meta-analysis. Dis Colon Rectum. 1995 Jul;38(7):687-94. doi: 10.1007/BF02048023. PMID 7607026
- [Derived] Salgueiro P, Garrido M, Santos RG, Pedroto I, Castro-Pocas FM. Polidocanol Foam Sclerotherapy Versus Rubber Band Ligation in Hemorrhoidal Disease Grades I/II/III: Randomized Trial. Dis Colon Rectum. 2022 Jul 1;65(7):e718-e727. doi: 10.1097/DCR.0000000000002117. Epub 2022 Nov 22. PMID 34840294